CLINICAL TRIAL: NCT05341102
Title: A Study to Evaluate the Safety and Pharmacokinetics of Single and Repeated Doses of CNTX-0290 in Healthy Subjects
Brief Title: A Study of Single and Repeated Doses of LY3556050 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: 18327; J2P-MC-LXBB (Other: Eli Lilly and Company)
Record Dates: First submitted 2022-04-18; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: All the participants will be double blinded except for LY3556050 (Part 1) - Cohort 7 which will be open label.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- LY3556050 (Part 1) (Experimental): Participants will receive single ascending doses of LY3556050 orally.
  Interventions: Drug: LY3556050
- Placebo (Part 1) (Experimental): Participants will receive placebo orally.
  Interventions: Drug: Placebo
- LY3556050 (Part 2) (Experimental): Participants will receive multiple ascending doses of LY3556050 orally.
  Interventions: Drug: LY3556050
- Placebo (Part 2) (Experimental): Participants will receive placebo orally.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3556050 — Administered orally.
  Other Names: CNTX-0290
  Arms: LY3556050 (Part 1); LY3556050 (Part 2)
Drug: Placebo — Administered orally.
  Arms: Placebo (Part 1); Placebo (Part 2)

SUMMARY:
The main purpose of this study is to conduct blood tests to measure how much LY3556050 is in the bloodstream and to determine if any age, gender, or food effects exist. The study will also evaluate the safety of LY3556050. This is a 2-part study. In Part 1, single increasing doses of LY3556050 will be given orally and participants will be confined for a 5-day period. In Part 2, multiple increasing doses of LY3556050 will be given orally and participants will be confined for a 14-day period.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation.
* Participants with a body mass index (BMI) of 18.0 to 35.0 kilograms per square meter (kg/m²) and have body weight of 50 kg or more.

Exclusion Criteria:

* Has any history of or active cardiac disease, including congestive heart failure, angina, any arrhythmia, or clinically significant findings on Electrocardiogram (ECG).
* Has diabetes mellitus, acromegaly, clinically active thyroid disease, or other active endocrinopathy.
* Has asthma or other severe respiratory disease.
* Is pregnant, lactating, or planning a pregnancy.
* Has active alcohol or substance abuse or history of alcohol or substance abuse within the 6 months prior to randomization.
* Any abnormal laboratory finding or vital signs outside specified parameters.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2017-06-02 (Actual); Study Completion 2017-06-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Event(s) (SAEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline through Day 30
  A summary of TEAEs, SAEs and other non-serious adverse events (AEs), regardless of causality, will be reported in the Reported Adverse Events module
Pharmacokinetics (PK): Maximum Concentration (Cmax) of LY3556050 (Part 1) | Predose on day 1 until Day 3 (Cohorts 1 to 7), and Predose on Day 8 until Day 10 (Only for Cohort 7)
  PK: Cmax of LY3556050 (Part 1)
PK: Area Under the Plasma Concentration Versus Time Curve From Zero to Infinity (AUC[0-∞]) of LY3556050 (Part 1) | Predose on day 1 until Day 3 (Cohorts 1 to 7), and Predose on Day 8 until Day 10 (Only for Cohort 7)
  PK: AUC[0-∞] of LY3556050 (Part 1)
PK: Fraction of LY3556050 Excreted in 48-hour Urine (fe[0-48]) (Part 1) | Predose on day 1 until Day 3 (Cohort 7), and Predose on Day 8 until Day 10 (Cohort 7)
  PK: fe[0-48] of LY3556050 (Part 1)
PK: Cmax of LY3556050 (Part 2) | Predose up to Postdose on Day 10
  PK: Cmax of LY3556050 (Part 2)
PK: Area Under the Plasma Concentration Versus Time Curve From Zero to 24 Hours (AUC[0-24]) of LY3556050 (Part 2) | Predose up to Postdose on Day 10
  PK: AUC[0-24] of LY3556050 (Part 2)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Medpace Clinical Pharmacology, LLC, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No